CLINICAL TRIAL: NCT01960595
Title: Comparison of the Efficacy and Cost Analysis of Regional Anesthesia and Intravenous Fentanyl for Postoperative Pain Management in Patients Undergoing Hullax Valgus Surgery
Brief Title: Post-operative Pain Management In Patients Undergoing Hullax Valgus Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUH-IRB-20120357
Record Dates: First submitted 2013-09-13; First posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-05

CONDITIONS: Pain
Keywords: PCA,Nerve block,Hullax Valgus
MeSH Terms: conditions — Pain | interventions — Nerve Block

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IV fentanyl PCA (Experimental): The patient receives post-OP IV fentanyl PCA
  Interventions: Procedure: IV fentanyl PCA
- post-OP IV fentanyl PCA and local infiltration (Active Comparator): pretreatment of local infiltration 0.25% bupivacaine 5 ml and post-OP IV fentanyl PCA
  Interventions: Procedure: local bupivacaine infiltration and post-OP IV fentanyl PCA
- nerves block and post-OP IV fentanyl PCA (Active Comparator): pretreatment of peroneal nerves 0.25% bupivacaine 10 ml and post-OP IV fentanyl PCA
  Interventions: Procedure: Nerve Blocks and post-OP IV fentanyl PCA

INTERVENTIONS:
Procedure: IV fentanyl PCA
  Arms: IV fentanyl PCA
Procedure: local bupivacaine infiltration and post-OP IV fentanyl PCA
  Arms: post-OP IV fentanyl PCA and local infiltration
Procedure: Nerve Blocks and post-OP IV fentanyl PCA
  Arms: nerves block and post-OP IV fentanyl PCA

SUMMARY:
The purpose of this study is to investigate the efficacy and cost analysis of intravenous fentanyl combined with either local anesthesia infiltration or peroneal nerves block in patients with Hallux Valgus undergoing orthopedic corrective surgery and compared with patients without local anesthetics administration perioperatively.

ELIGIBILITY:
Inclusion Criteria:

1. patients with American Society of Anesthesiologists physical status I-III
2. aged 20-65 years
3. Requiring local anesthesia and PCA use
4. No severe cardiac or pulmonary diseases
5. BMI <35 kg/m2

Exclusion Criteria:

1. BMI ≧35 kg/m2
2. age > 65years
3. allergy to opioid or local anesthetics

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-02 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
provides adequate pain relief and decreases fentanyl consumption | including of surgery and 36 hours after surgery
  Patients are subgrouping into groups of post-OP IV fentanyl PCA only, pretreatment of local bupivacaine infiltration and post-OP IV fentanyl PCA, and pretreatment of peroneal nerves block and post-OP IV fentanyl PCA. Resting pain and moving pain scores are measured by the numeric rating scale and classified into none, mild, moderate and severe pain four grades. Pains scale and side effects are recorded at time intervals of post-OP 0 hours, 6 hours, 12 hours, 24 hours, and 36 hours after surgery.

SECONDARY OUTCOMES:
incidence of side effects and complications | intraoperatively and 36 hours after surgery
  side effects include of intraoperative hypo-tension,dizziness, nausea, and vomiting.

OTHER OUTCOMES:
assessment of cost analysis among groups | surgery period and 36 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Peng Ju Huang, MD, PhD., Study Director — Department of orthopaedic surgery, Kaohsiung Medical University, Taiwan
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung, Taiwan